CLINICAL TRIAL: NCT04057833
Title: A Phase 1 Open-Label, Single-Center Investigator Initiated Trial (IIT) of E-CEL UVEC Cells as an Adjunct Cell Therapy for the Arthroscopic Rotator Cuff Repair in Adults
Brief Title: E-CEL UVEC Cells as an Adjunct Cell Therapy for the Arthroscopic Rotator Cuff Repair in Adults
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Angiocrine Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0809
Record Dates: First submitted 2019-07-30; First posted 2019-08-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tears; Muscle Atrophy or Weakness; Tendon Rupture - Shoulder; Safety Issues
Keywords: Cell Therapy; Supraspinatus tendon; Systemic safety and toxicity; Muscle and Tendon quality
MeSH Terms: conditions — Rotator Cuff Injuries; Muscular Atrophy; Asthenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E-CEL UVEC (Experimental): Patients will receive an injection of the Cell therapy vehicle into their supraspinatus muscle and tendon at the time of rotator cuff repair.
  E-CEL UVEC cells suspended in autologous plasma and combined with thrombin at the implantation site (tendon delivery).
  E-CEL UVEC cells suspended in 6.0% Dextran 40 and 10.0% human serum albumin (HSA) (infusion solution) (muscle delivery).
  Interventions: Drug: E-CEL UVEC

INTERVENTIONS:
Drug: E-CEL UVEC — Local implantation of E-CEL UVEC cells at the supraspinatus tendon repair site

SUMMARY:
This is a phase 1b investigator-initiated clinical trial that will evaluate the safety and feasibility of E-CEL UVEC® cells with the aim of improving outcomes for patients with full-thickness rotator cuff tears who undergo arthroscopic surgical repair.

Allogeneic E-CEL UVEC cells will be delivered to the tendon repair site and to the muscle adjacent to the tendon repair site.

DETAILED DESCRIPTION:
Full-thickness rotator cuff tears present a clinical challenge, often with occurrence of re-tears after surgical repair and a slow rate of complete functional recovery, which limits daily functional tasks and has negative impacts on qualify-of-life. The frequency of failed healing and re-tear following repair is more pronounced in patients over age 60 due to age-related, intrinsic degenerative changes involving the muscle, tendon, and enthesis.

Healing of the enthesis, the site of tendon attachment to the bone, can be compromised due to microvascular and vascular niche deficiencies resulting from various causes including aging, prior injuries, and/or tissue degeneration.

There is currently no approved adjunct biologic therapy to improve surgical repairs of full rotator cuff tear, enhance post-operative recovery, and decrease the risk of re-tear. This trial will investigate the safety and feasibility of local implantation of E-CEL UVEC cells along with standard-of-care arthroscopic surgical repair of full rotator cuff tears. E-CEL UVEC cells are proprietary allogeneic human umbilical vein endothelial cells produced under cGMP and cGTP regulations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45-70 years old
* Diagnosis of full-thickness supraspinatus tendon tear by MRI and physical examination
* Tendon retraction 1 to 3 cm on MRI
* Goutallier score ≤ grade 2.
* Failed standard non-operative treatments for tendon tear including a minimum of 3 months of physical therapy as well as oral anti-inflammatory medications, subacromial steroid injection, activity modification, etc.

Exclusion Criteria:

* Tears of any cuff tendon other than the supraspinatus
* Frank signs of glenohumeral osteoarthritis on MRI
* Diagnosis of acute tendon tear
* Lack of significant pain and/or loss of function due to tendon tear History of previous rotator cuff repair
* History of upper extremity fracture or other moderate to severe upper extremity trauma
* BMI < 20 or > 35
* Diagnosis of Type I or type II diabetes, or other metabolic disorders
* Previous history of cancer. Subjects with cervical carcinoma in situ or localized basal or squamous cell carcinoma treated with definitive surgery are eligible.
* Diagnosis of an autoimmune disorder Know history of HIV
* Current use of nicotine products
* History of diabetes, malignancy within 5 years of the procedure, immunosuppression, autoimmune or connective tissue disorders such as lupus or rheumatoid arthritis, schizophrenia or other psychiatric disorder that could interfere with postoperative rehabilitation, or other disability that would obviously adversely impact the patient's ability to participate in standard postoperative rehabilitation
* Pregnancy
* Inability to comply with post-operative rehabilitation
* Hypersensitivity reactions to bovine (cow) proteins

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Short-term safety | 0 surgery to +11 days post op
  The primary study outcomes are measures of local and systemic safety and toxicity via adverse event (AE) logs (post-operative day 0 to Day 11). AE are evaluated using a 5 point severity scale to grade the AE, 1 (mild) to 5 (death/ fatal).

SECONDARY OUTCOMES:
Long-term safety | post-operative 90 day to 1 year following the surgical repair
  The primary study outcomes are measures of local and systemic safety and toxicity via symptom reporting (post-operative day +90 to 1 year post-op). Symptom reporting will evaluate pain and swelling based on a 0 to 100mm visual analog scale range, in addition to further symptom reporting.
MRI | post-operative 90 day to 1 year
  Re-tear rate based on clinical and MRI evaluation for MRI assessments of muscle and tendon quality, measured as a percentage of total volume (%).
Strength | post-operative 90 day to 1 year
  Shoulder strength during regular intervals post-operatively up to 1 year. BioDex system 3 will measure Peak Toque in Nm, scapular plane abduction strength 0-90 degrees.
PROMS | post-operative 90 day to 1 year
  Patient-reported outcomes post-operatively up to 1 year. ASES affected vs unaffected shoulder score (each test has a maximum score of 100 points).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rodeo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Voigt C, Bosse C, Vosshenrich R, Schulz AP, Lill H. Arthroscopic supraspinatus tendon repair with suture-bridging technique: functional outcome and magnetic resonance imaging. Am J Sports Med. 2010 May;38(5):983-91. doi: 10.1177/0363546509359063. PMID 20436053
- [Background] Ippolito E, Natali PG, Postacchini F, Accinni L, De Martino C. Morphological, immunochemical, and biochemical study of rabbit achilles tendon at various ages. J Bone Joint Surg Am. 1980;62(4):583-98. PMID 6991502
- [Background] Tempfer H, Traweger A. Tendon Vasculature in Health and Disease. Front Physiol. 2015 Nov 18;6:330. doi: 10.3389/fphys.2015.00330. eCollection 2015. PMID 26635616
- [Background] Hein J, Reilly JM, Chae J, Maerz T, Anderson K. Retear Rates After Arthroscopic Single-Row, Double-Row, and Suture Bridge Rotator Cuff Repair at a Minimum of 1 Year of Imaging Follow-up: A Systematic Review. Arthroscopy. 2015 Nov;31(11):2274-81. doi: 10.1016/j.arthro.2015.06.004. Epub 2015 Jul 15. PMID 26188783
- [Background] Rodeo SA. Biologic augmentation of rotator cuff tendon repair. J Shoulder Elbow Surg. 2007 Sep-Oct;16(5 Suppl):S191-7. doi: 10.1016/j.jse.2007.03.012. Epub 2007 Jun 15. PMID 17574875
- [Background] Butler JM, Gars EJ, James DJ, Nolan DJ, Scandura JM, Rafii S. Development of a vascular niche platform for expansion of repopulating human cord blood stem and progenitor cells. Blood. 2012 Aug 9;120(6):1344-7. doi: 10.1182/blood-2011-12-398115. Epub 2012 Jun 18. PMID 22709690
- [Background] Ding BS, Nolan DJ, Butler JM, James D, Babazadeh AO, Rosenwaks Z, Mittal V, Kobayashi H, Shido K, Lyden D, Sato TN, Rabbany SY, Rafii S. Inductive angiocrine signals from sinusoidal endothelium are required for liver regeneration. Nature. 2010 Nov 11;468(7321):310-5. doi: 10.1038/nature09493. PMID 21068842
- [Background] Ding BS, Nolan DJ, Guo P, Babazadeh AO, Cao Z, Rosenwaks Z, Crystal RG, Simons M, Sato TN, Worgall S, Shido K, Rabbany SY, Rafii S. Endothelial-derived angiocrine signals induce and sustain regenerative lung alveolarization. Cell. 2011 Oct 28;147(3):539-53. doi: 10.1016/j.cell.2011.10.003. PMID 22036563
- [Background] Candotti F, Shaw KL, Muul L, Carbonaro D, Sokolic R, Choi C, Schurman SH, Garabedian E, Kesserwan C, Jagadeesh GJ, Fu PY, Gschweng E, Cooper A, Tisdale JF, Weinberg KI, Crooks GM, Kapoor N, Shah A, Abdel-Azim H, Yu XJ, Smogorzewska M, Wayne AS, Rosenblatt HM, Davis CM, Hanson C, Rishi RG, Wang X, Gjertson D, Yang OO, Balamurugan A, Bauer G, Ireland JA, Engel BC, Podsakoff GM, Hershfield MS, Blaese RM, Parkman R, Kohn DB. Gene therapy for adenosine deaminase-deficient severe combined immune deficiency: clinical comparison of retroviral vectors and treatment plans. Blood. 2012 Nov 1;120(18):3635-46. doi: 10.1182/blood-2012-02-400937. Epub 2012 Sep 11. PMID 22968453
- [Background] Gori JL, Butler JM, Kunar B, Poulos MG, Ginsberg M, Nolan DJ, Norgaard ZK, Adair JE, Rafii S, Kiem HP. Endothelial Cells Promote Expansion of Long-Term Engrafting Marrow Hematopoietic Stem and Progenitor Cells in Primates. Stem Cells Transl Med. 2017 Mar;6(3):864-876. doi: 10.5966/sctm.2016-0240. Epub 2016 Oct 14. PMID 28297579
- [Background] Poulos MG, Ramalingam P, Gutkin MC, Llanos P, Gilleran K, Rabbany SY, Butler JM. Endothelial transplantation rejuvenates aged hematopoietic stem cell function. J Clin Invest. 2017 Nov 1;127(11):4163-4178. doi: 10.1172/JCI93940. Epub 2017 Oct 16. PMID 29035282
- [Background] Poulos MG, Crowley MJP, Gutkin MC, Ramalingam P, Schachterle W, Thomas JL, Elemento O, Butler JM. Vascular Platform to Define Hematopoietic Stem Cell Factors and Enhance Regenerative Hematopoiesis. Stem Cell Reports. 2015 Nov 10;5(5):881-894. doi: 10.1016/j.stemcr.2015.08.018. Epub 2015 Oct 1. PMID 26441307
- [Background] Potter HG, Linklater JM, Allen AA, Hannafin JA, Haas SB. Magnetic resonance imaging of articular cartilage in the knee. An evaluation with use of fast-spin-echo imaging. J Bone Joint Surg Am. 1998 Sep;80(9):1276-84. doi: 10.2106/00004623-199809000-00005. PMID 9759811
- [Background] Koff MF, Pownder SL, Shah PH, Yang LW, Potter HG. Ultrashort echo imaging of cyclically loaded rabbit patellar tendon. J Biomech. 2014 Oct 17;47(13):3428-32. doi: 10.1016/j.jbiomech.2014.08.018. Epub 2014 Sep 1. PMID 25234349